CLINICAL TRIAL: NCT01372254
Title: Behavioral Intervention for Low Income Depressed Smokers in Drug Treatment
Acronym: BA-DAS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Laura MacPherson, Dr. Laura MacPherson, University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RSGT1101101CPPD
Record Dates: First submitted 2011-06-10; First posted 2011-06-13 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Cigarette Smoking; Drug Use
Keywords: Cigarette Smoking; Drug Use; Depressed Mood
MeSH Terms: conditions — Cigarette Smoking; Consciousness Disorders | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard smoking cessation (Active Comparator): Participants will receive a standard smoking cessation treatment in individual format. Treatment will be delivered in five, 90-minute individual sessions, and with two booster sessions assessed scheduled 2 and 4 weeks post quit. Participants will also receive 8 weeks of the transdermal nicotine patch.
  Interventions: Behavioral: Standard Treatment; Drug: Transdermal Nicotine Patch
- BA for substance abusing smokers (Experimental): The Behavioral Activation for Drug Abusing Smokers (BA-DAS) treatment protocol will incorporate elements of the ST along with behavioral activation strategies, modified for smoking. Treatment will consist of five, 90-minute individual sessions, and with two booster sessions scheduled 2 and 4 weeks post quit. Participants will also receive 8 weeks of the transdermal nicotine patch.
  Interventions: Behavioral: BAD-AS; Drug: Transdermal Nicotine Patch

INTERVENTIONS:
Behavioral: Standard Treatment — Participants will receive a standard smoking cessation treatment in individual format. Treatment will be delivered in five, 90-minute individual sessions, and with two booster sessions assessed scheduled 2 and 4 weeks post quit. Participants will also receive 8 weeks of the transdermal nicotine patch.
  Other Names: ST
  Arms: Standard smoking cessation
Behavioral: BAD-AS — The Behavioral Activation for Drug Abusing Smokers (BA-DAS) treatment protocol will incorporate elements of the ST along with behavioral activation strategies, modified for smoking. Treatment will consist of five, 90-minute individual sessions, and with two booster sessions scheduled 2 and 4 weeks post quit. Participants will also receive 8 weeks of the transdermal nicotine patch.
  Arms: BA for substance abusing smokers
Drug: Transdermal Nicotine Patch — 8 weeks of the Transdermal Nicotine Patch Nicoderm CQ at 24 hour doses of 21, 14, and 7 mg respectively depending on participant's initial level of nicotine use. Nicotine patch dose will decrease at 2 or 4 week increments also specific to the participant's initial nicotine level. Participants in both intervention arms will receive transdermal nicotine patch.
  Other Names: Nicoderm CQ

SUMMARY:
The objective of the proposed project is to develop a novel, behavioral approach to smoking cessation that can be integrated with residential drug use treatment for low income substance using smokers with elevated depressive symptoms. The approach utilizes behavioral activation strategies which have been shown to reduce smoking among community samples and which can be easily targeted for the particular needs of low income substance users.

DETAILED DESCRIPTION:
This project will take place in two phases. In the first phase, the investigators will utilize pilot testing with 10 participants (two groups of 5 individuals) to integrate two existing behavioral activation manuals to develop the Behavioral Activation for Drug Abusing Smokers (BA-DAS). In Phase II, the investigators will randomize 80 patients to either: 1) standard smoking cessation treatment (ST) and nicotine replacement therapy (NRT) or 2) BA-DAS (which includes ST and NRT). Based on the outcome of this preliminary trial, the BA-DAS protocol will be further refined and readied for larger-scale clinical trials to develop a comprehensive approach to treating smoking among low income, largely minority, depressed smokers in residential drug use treatment, which may be instrumental in reducing smoking among this especially at risk group.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 years of age
* regular smoker for at least one year
* currently smoking an average ≥ 10 cigarettes (also cigarellos, bidis, or Black and Milds included) per day
* report motivation to quit smoking in the next month
* report elevated depressive symptoms

Exclusion Criteria:

* physical concerns contraindicating the nicotine patch
* limited mental competency and/or the inability to give informed, voluntary, written consent to participate
* current use of pharmacotherapy for smoking cessation not provided by the researchers during the quit attempt
* use of psychotropic medication for < 3 months
* primary use of other tobacco products (specifically: chewing tobacco, cigars, and pipes)
* psychotic symptoms
* current pregnancy or plans to become pregnant within the following three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura MacPherson, PhD, Principal Investigator — University of Maryland
Locations (1):
- Salvation Army Harbor Light Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Smoking Cessation | BA for Substance Abusing Smokers
Started | 47 | 49
Completed | 43 | 46
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Population: Analysis population is not different from the assignment in Participant Flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Smoking Cessation | BA for Substance Abusing Smokers | Total
Number analyzed (Participants) | 47 | 49 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 49 | 94
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.98 (9.69) | 42.57 (10.58) | 43.25 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 32 | 33 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 42 | 47 | 89
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 47 | 49 | 96

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Smoking-Abstinent for 7 Days, 26 Weeks Post Quit Date
Description: 7 days of smoking abstinence confirmed biochemically at 26 weeks
Time Frame: 26 weeks post quit date
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Smoking Cessation | BA for Substance Abusing Smokers
Number analyzed (Participants) | 47 | 49
Participants | 5 | 1

ADVERSE EVENTS:
Time Frame: 3 years, 3 months. Adverse events were monitored through study completion.
Description: Definition of adverse event/or serious adverse event does not differ from clinicaltrials.gov definitions.
Arm/Group | Standard Smoking Cessation | BA for Substance Abusing Smokers
All-Cause Mortality (participants affected / at risk) | 1/47 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/49
Other Adverse Events (participants affected / at risk) | 0/47 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No